CLINICAL TRIAL: NCT06370546
Title: Evaluation of Cardiac Response to High and Low-Intensity Strength Training in Hypertensive Subjects
Brief Title: Cardiac Response to Strength Training in Hypertensive Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Católica del Maule (Other)
Responsible Party: Principal Investigator, Antonio Roberto Zamunér, Adjunct Professor, Universidad Católica del Maule
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 229/2022
Record Dates: First submitted 2024-04-12; First posted 2024-04-17 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Physical Exercise; Hypertension
MeSH Terms: conditions — Motor Activity; Hypertension | interventions — Ultrasonic Waves

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial, single blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Low Intensity (Experimental): The low-intensity group undergoes a strength training program using barbells, weights and dumbbells, consisting of 6 sets of 12 repetitions each, with an execution speed below 40% of the maximum velocity used in the one-repetition maximum
  Interventions: Other: Low intensity
- high intensity (Experimental): The low-intensity group undergoes a strength training program using barbells, weights and dumbbells consisting of 6 sets of 6 repetitions each, with an execution speed equal to or greater than 80% of the maximum velocity used in the one-repetition maximum
  Interventions: Other: high intensity

INTERVENTIONS:
Other: Low intensity — Low intensity group: participants will be requested to perform the following exercises: 1)squat, 2) rowing, 3)deadlift and 4)bench press. All exercises will be performed with low intensity (40% of the maximum velocity used in one-repetition maximum) and will be supervised by a researcher.
  Arms: Low Intensity
Other: high intensity — High intensity group: participants will be requested to perform the following exercises: 1)squat, 2)rowing, 3)deadlift and 4)bench press. All exercises will be performed with high intensity (80% of the maximum velocity used in one-repetition maximum) and will be supervised by a researcher.
  Arms: high intensity

SUMMARY:
This study aims to determine the acute effects of high and low-intensity strength training on cardiac autonomic control in hypertensive subjects

DETAILED DESCRIPTION:
The present study aims to determine the cardiovascular response in hypertensive individuals between 30 and 60 years old to one session of high and low intensity strength training.

Participants will undergo a low-intensity strength training including squats, barbell rows, deadlifts and chest presses with a load dynamic of 12 repetitions for 6 sets at an execution speed of less than 55 % of your maximum weight. This is followed by a one-week washout period. Subsequently, high intensity strength training is performed with the same exercises but with a load of 6 repetitions for 6 series at an intensity greater than 80% of the maximum repetition speed. The order of the sessions will be random.

After each session, blood pressure will be recorded for 24 hours using a holter monitor, which will report pressures during both day and night

The results obtained will be determined by the differences in the before and after values. Consequently, the behavior of the following variables: 1) heart rate variability, 2) blood pressure and 3) heart rate will determine the final results of this research.

The entire study will be carried out at the Catholic University of Maule, in its Kinesiology laboratory.

ELIGIBILITY:
Inclusion Criteria:

* Participants exclusively diagnosed with hypertension by a medical professional

Exclusion Criteria:

* Participants with any other chronic medical condition
* Subjects with any upper or lower limb injury that prevents strength training
* Subjects with cardiovascular abnormalities other than hypertension

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2023-03-20 (Actual); Primary Completion 2024-07-20 (Actual); Study Completion 2024-07-20 (Actual)

PRIMARY OUTCOMES:
Heart rate variability | 2 hours
  Determine the effects of high and low-intensity strength training on heart rate variability, based on the time between each heartbeat, during the assessment
Blood pressure systolic | 24 hours
  Determine the effects of high and low intensity resistance training on blood pressure with a blood pressure monitor for 24 hours.
Blood pressure diastolic | 24 hours
  Determine the effects of high and low intensity resistance training on blood pressure diastolic with a blood pressure monitor for 24 hours.
Blood pressure mean | 24 hours
  Determine the effects of high and low intensity resistance training on blood pressure mean with a blood pressure monitor for 24 hours.
Heart Rate | 24 hours
  Determine the effects of high and low intensity strength training on the behavior of heart rate, using a heart rate monitor, throughout the intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Católica del Maule, Talca, Maule Region, Chile